CLINICAL TRIAL: NCT00334165
Title: Auricular Acupuncture (AA) vs. Sham Acupuncture for Complementary Analgesia During Elective Total Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: Auricular Acupuncture for Analgesia During Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Humboldt-Universität zu Berlin (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: III UV 13/05
Record Dates: First submitted 2006-06-03; First posted 2006-06-06 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Acute Pain; Total Hip Arthroplasty
MeSH Terms: conditions — Acute Pain | interventions — Acupuncture, Ear

INTERVENTIONS:
Procedure: Auricular acupuncture (procedure)

SUMMARY:
The aim is to investigate whether auricular acupuncture is superior to sham acupuncture in relief of acute pain and in reduction of analgesics in patients during total hip arthroplasty

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an American Society of Anesthesiologists physical status of I to III scheduled for elective hip arthroplasty because of degenerative osteoarthritis under general anesthesia.
2. Surgery time does not exceed 100 minutes.
3. Patients without previous opioid medication.
4. Patients ranged 45-85 years old.
5. Patients who have given informed consent.

Exclusion Criteria:

1. Pregnant or nursing females.
2. Recidivist alcoholics.
3. Local or systemic infection.
4. Age < 45 and > 85 years.
5. Surgery time more than 100 minutes.
6. Intraoperative complications (bleeding, required blood transfusion more than 4 units of packed cells , cardiovascular instability, required catecholamines).
7. Patients consumed opioid medication before surgery.
8. Patients with prosthetic or damaged cardiac valves.
9. Patients who are unable to understand the consent form.
10. History of psychiatric disease.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2008-06

PRIMARY OUTCOMES:
Intraoperative analgesics requirement

CONTACTS AND LOCATIONS:
Overall Officials: Taras I Usichenko, M.D., Study Chair — Ernst Moritz Arndt University
Locations (2):
- Germany (2):
  - University of Berlin, Campus Charite, Berlin
  - Ernst Moritz Arndt University, Greifswald